CLINICAL TRIAL: NCT04041258
Title: "Evaluation of Clinical and Radiographic Results of Pseudarthrosis of Clavicle Treated With Plaque and Screws"
Acronym: CLAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the number of patients was not sufficient to support continuation of the study
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAPS
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-08

CONDITIONS: Pseudoarthrosis of the Clavicle
Keywords: pseudoarthrosis; clavicle
MeSH Terms: conditions — Clavicle, Pseudarthrosis Of, Congenital; Pseudarthrosis

STUDY DESIGN:
Intervention Model Description: interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- evaluation of clinical and radiographic findings after surgical treatment (Experimental): Evaluation of clinical and radiographic findings at least 1 year after surgical treatment for pseudoarthrosis of clavicle
  Interventions: Procedure: pseudoarthrosis of clavicle

INTERVENTIONS:
Procedure: pseudoarthrosis of clavicle — Pseudoarthrosis represents a complication following a fracture, resulting in persistent symptoms and functional limitation, which prolongs the recovery time for the patient and necessitates new surgery. The purpose of surgery for pseudoarthrosis is to re-establish the length and alignment of the clavicle in an environment favorable to the union of bone fragments.

SUMMARY:
This is an interventional study for clinical and radiographic evaluation of patients operated for pseudoarthrosis of the clavicle

DETAILED DESCRIPTION:
The aim of our study is to collect clinical and radiographic data from patients operated for pseudoarthrosis of the clavicle from 2007 to 2017 at the Rizzoli Orthopedic Institute, in order to evaluate the clinical and radiographic results of the treatment. This is an interventional study and patients will be contacted by telephone to verify their willingness to perform a visit (including a bilateral radiographic) at the Rizzoli Orthopedic Institute

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of pseudarthrosis intervention
2. Males and Females
3. Patients treated for pseudoarthrosis of the clavicle between 2007 and 2017 at the Rizzoli Orthopedic Institute

Exclusion Criteria:

1. Floating shoulder
2. subjects who present contraindications to radiographic examination at the time of telephone contact

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
range of motion ROM | at least 1 year of follow up
  improvement of range of motion measure (in grade)
presence of dyskinesias | at least 1 year of follow up
  objective clinical evaluation (elevation, external rotation, abduction) with constant scale (0-25 points)
alteration of the clavicle length | at least 1 year of follow up
  measure (mm) obtained from radiographic evaluation

SECONDARY OUTCOMES:
evaluate shoulder function | at least 1 year of follow up
  improvement in Assessment Shoulder and Elbow Scale (ASES) (0-100 points)

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No